CLINICAL TRIAL: NCT06429397
Title: A Single-arm, Multicenter, Prospective Phase II Clinical Study of Anlotinib Combined With Benmelstobart in the First-line Treatment of Advanced Pheochromocytoma/Paraganglioma
Brief Title: Anlotinib Combined With Benmelstobart for Advanced Pheochromocytoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-304
Record Dates: First submitted 2024-04-08; First posted 2024-05-28 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pheochromocytoma
MeSH Terms: conditions — Pheochromocytoma | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug (Experimental): Patients receive Penpulimab and anlotinib
  Interventions: Drug: Anlotinib and Benmelstobart

INTERVENTIONS:
Drug: Anlotinib and Benmelstobart — Enrolled patients received a treatment cycle every 21 days: 200mg of piamprizumab was given intravenously on the first day of treatment, and 12mg of anrotinib hydrochloride capsule was given continuously for 14 days and suspended for 7 days.

SUMMARY:
There is currently no standard first-line treatment for stage PPGL, and the 5-year survival rate of patients with advanced pheochromocytoma/paraganglioma (PPGL) is low, ranging from 30% to 60%. At present, several domestic teams have carried out clinical studies on the treatment of advanced PPGL with good efficacy. In the early stage, our center used anrotinib to treat advanced PPGL, and the overall effective rate reached 44%. In the early stage, our team used anrotinib combined with PD-1 monoclonal antibody to treat advanced PPGL patients. The effective rate reached 66% (2/3). Therefore, the investigators plan to further conduct prospective studies to explore the efficacy and safety of anlotinib combined with PD-1 monoclonal antibody in the treatment of advanced PPGL, so as to bring benefits to patients with advanced PPGL.

DETAILED DESCRIPTION:
1.1 Adrenal pheochromocytoma/paraganglioma pheochromocytoma (PCC) and Paraganglioma (PGL) (pheochromocytoma and paraganglioma (PPGL) are rare malignant tumors with neuroendocrine function and metastatic potential. The incidence is 0.4-2.1 persons/million, 80%-85% originate from the adrenal medulla, and 15%-20% originate from the neural crest tissue from the neck to the pelvis. The PPGL metastasis rate at initial diagnosis is 10%, and the risk of metastasis is as high as 34-69% for those with SDHB gene mutations. The recurrence rate of PPGL patients after radical resection was 30%, 47% recurred with multiple nodules, 58% with metastasis. The most common sites of metastasis were lymph nodes and bone (70-80%), followed by lung and liver (50%). In addition, some PPGL is difficult/unresectable due to its proximity to important structures such as large blood vessels or nerves, and the 5-year survival rate for advanced PPGL is 30%-60%.

Early PPGL can be cured by surgery, but late PPGL is mainly systemic therapy, such as chemotherapy, targeted drugs and nuclide therapy. The main chemotherapy regimen for advanced PPGL is cyclophosphamide - vincristine - dacarbazine (CVD regimen), and ESMO guidelines recommend CVD for patients with rapid tumor progression and heavy tumor burden. The objective response rate of CVD regimen was 33%, the median duration of response was 1.3 years, and the 5-year survival rate of patients with effective CVD was 51%. The main limitations of CVD in the treatment of advanced PPGL are (1) The average number of cycles required for CVD chemotherapy is 11.6±10.8 months; (2) The incidence of CVD related toxicity, such as bone marrow suppression and neurotoxicity, was 50%. Some patients could not maintain treatment due to intolerance, and long-term use of the above drugs could increase the incidence of hematological tumors, which may be related to the alkylating properties of daparbazine.

Domestic guidelines and the FDA recommend 131I-MIBG for the treatment of advanced PPGL. Loh et al. reviewed and analyzed 21 central LSA-131I-MIBG clinical studies: 30% patients could have Partial Response (PR); Gonias S et al. Phase II clinical study of HSA-131I-MIBG in the treatment of advanced PPGL: 22% of patients could have PR. Two 131I-MIBGs show good efficacy, but there are no phase III clinical studies to further validate efficacy and safety. Limitations of radionuclide therapy lie in (1) the narrow range of indications: (1) ESMO guidelines indicate that only 50% of patients with positive MIBG scan are suitable. ② Pregnant women and pregnant patients should not use; (2) Severe hematological toxicity: the incidence of myosuppression was 4%-79%, about 40% of patients treated with low-dose 131I-MIBG had grade 3/4 toxicity, while those treated with high-dose 131I-MIBG had up to 80%, of which 25% needed hematological therapy and secondary hematological tumors could be developed . (3) Hypogonadism. In addition, at present, the units that can carry out nuclide therapy in China are limited, and patients can not perform nuclide therapy again after receiving progress of nuclide therapy.

1.2 Tyrosine kinase inhibitors (TKI) and advanced adrenal pheochromocytoma/paraganglioma Tyrosine kinase (TK) is a key site in the activation and regulation of cell proliferation signaling pathways. Abnormal TK pathway caused by mutation, translocation or amplification can lead to tumor occurrence, progression, invasion and metastasis. Tyrosine kinase inhibitors (TKI) mainly act on vascular endothelial growth factor receptor (VEGFR), platelet growth factor (PDGFR) and insulin family receptor (InsR). TKI acts on advanced PPGL through the pseudo-hypoxia pathway and VEGF angiogenesis pathway.

Advanced PPGL with abundant blood supply and high expression of angiogenic factor (VEGF) can promote tumor neovascularization and provide oxygen and nutrition for tumors. TKI has a good therapeutic effect on advanced PPGL with high VEGF expression, which may be related to its blocking of VEGF signaling pathway, continuous inhibition of tumor neovascugenesis and promotion of abnormal blood vessel normalization. In addition, HIF axis misalignment can also promote the development and transfer of PPGL. SDH gene mutations are the most common in PPGL (including SDHA, SDHB, SDHC, SDHD), which cause abnormalities in the subunit encoding the succinate dehydrogenase complex (SDH) and block the tricarboxylic acid cycle (TCA). Abnormal TCA can inhibit hypoxia-inducing factor (HIF-α) proline hydroxylase, and HIF-α accumulation will activate the pseudo-hypoxia pathway and up-regulate the expression of VEGF and other factors.

ESMO guidelines recommend sunitinib for the treatment of advanced PPGL. Currently, the only prospective phase II clinical study showed that 3 cases (13%) had PR (SDHB, SDHD, RET gene mutations, respectively). A retrospective study of 17 cases of advanced PPGL treated by MD Anderson and Gustavvy-Roussy et al. showed that there were 3 cases of PR and 5 cases of SD (6 of which were SDHB or VHL gene mutations). In the study , grade 1-2 toxicity was the most common, with about 68% of patients presenting symptoms such as fatigue, nausea and vomiting, palm-plantar dyspepsia, etc., while only 56%/12% of patients presented 3/4 toxicity, mainly manifested as nausea, vomiting and hypertension, without hematological toxicity.

Retrospective studies have also shown that Renvastinib, pazopanib, acitinib and other TKI have certain efficacy in advanced PPGL, but there is a lack of prospective clinical evidence. Hassan Nelson L et al. treated 11 cases of advanced PPGL with lenvatinib, and the results were 5 cases PR, 3 cases SD, and the median PFS was 14.7 months. Mauricio Emmanuel Burotto Pichun et al. are conducting a study on the treatment of 11 cases of advanced PPGL with acitinib: 4 cases of PR and 6 cases of SD. The above studies show the preliminary efficacy of various TKI, and the effect may be better for SDHB mutations, with a controllable safety, mainly hypertension. In 2017, preliminary results of a prospective clinical study of cabotinib in the treatment of advanced PPGL were reported in the conference abstract: ORR of 45%, PFS of 11 months, and no grade 3/4 toxicity. In summary, TKI monotherapy in the treatment of advanced PPGL shows some effect, but it is still not satisfactory.

There is currently no standard first-line treatment for advanced PPGL. NCCN guidelines and China's expert consensus (2020 edition) recommend the use of tumor reduction surgery (palliative resection) combined with radiotherapy, radionuclide therapy or systemic chemotherapy and other treatment options, but the above methods have uncertain efficacy and certain limitations, still need to be confirmed by prospective experiments, so patients are recommended to participate in clinical trials.

1.3 Application of antirotinib hydrochloride in advanced adrenal pheochromocytoma/paraganglioma Allotinib (AL3818) is manufactured by Zhengda Tianqing Pharmaceutical Group Co., LTD. (CTTQ; Lianyungang, Jiangsu, China) self-developed TKI drugs, targeting VEGFR1-3, FGFR1-4, PDGFRα, G, β, rearrangement (RET) and stem cell factor receptor (c-Kit) during transfection [26]; Anlotinib has shown good anticancer activity in vitro/in vitro [27]. A multicentre, randomized, controlled Phase II clinical study of anlotinib in first-line treatment of metastatic renal cell carcinoma (mRCC) (NCT02072031)[28] showed similar efficacy of anlotinib and Sunitinib: There were no significant differences in median PFS (17.May vs. 16.June, P > 0.05), OS, ORR and DCR (P > 0.05), but the toxicity of anrotinib was lower, and the incidence of ≥3/4 toxicity was significantly lower than that of Sunitinib (28.9% vs.55.8%, P < 0.01). The main symptoms were hypertension and hand-foot syndrome, and no hematological toxicity was found. In addition, Lin J et al. also confirmed that anlotinib and Sunitinib had similar efficacy but higher safety. TKI treatment of advanced PPGL has a similar mechanism of action, but anlotinib safety may be better. In addition, our team has a certain foundation in the study of anrotinib in the treatment of advanced PPGL. In the early stage, anrotinib monotherapy was used to treat advanced PPGL in 4 cases and PR in 2 cases (1 case was a SHDB mutation), and the adverse reactions were mostly grade 1-2, with hypertension and hand-foot syndrome as the main manifestations. Therefore, antirotinib may have better efficacy and safety in advanced PPGL, which is worthy of further clinical exploration.

1.4 PD-1/PD-L1 monoclonal antibody kills tumors by activating its own normal anti-tumor immune mechanism. In 2014, Pembrolizumab achieved results in melanoma, officially ushering in the era of global immunotherapy. Subsequently, indications and significant curative effects were also obtained in multi-tumor species such as non-small cell lung cancer, gastric cancer and kidney cancer.

PD-L1 is mainly expressed in tumor cells and antigen-presenting cells (APCs), and is closely related to tumor immune escape [33] : PD-L1 receptor of tumor cell membrane binds to PD-1 receptor of T cell membrane, which weakens the ability of cytotoxic T lymphocytes to kill tumor cells. PD-1/PD-L1 mab blocks the above signaling process and restores/activates the anti-tumor activity of T cells.

A study in Peking Union Medical College Hospital [35] showed that 59.7% were positive for PPGL PD-L1 expression (HIS>10), and the positive rate of PD-L1 in advanced PPGL was 100%(1/1). Study [36] showed that PD-L1 expression was positive in 4 out of 10 advanced PPGL cases (40%). Studies indicated that the cytotoxic T lymphocyte infiltration level was increased in advanced PPGL (P=0.092). Therefore, PD-1 monoclonal antibody may have some significance in the treatment of advanced PPGL. At present, only A few cases have been reported in the treatment of advanced PPGL with PD-1 monoclonal antibody. The Phase II clinical study conducted by Naing A et al. in the treatment of advanced PPGL patients with pembrolizumab showed that 43% (4 cases) had no progress at 27 weeks (6.75 months). This suggests that PD-1 monoclonal antibody has a certain effect in the treatment of advanced PPGL, but PD-1 monotherapy can not meet the clinical needs.

KATO Y et al. proposed that the effective rate of PD-1 monoclonal antibody in the single treatment of solid tumors was 20%-30%, and the therapeutic effect was not satisfactory. The study of PD-1 monoclonal antibody combined with TKI in the treatment of liver cancer suggests that the combination of PD-1 monoclonal antibody can reverse the immunosuppressor tumor microenvironment in which PD-1 monoclonal antibody is ineffective, and assist PD-1/PD-L1 monoclonal antibody to activate cytotoxic T lymphocytes. The efficacy of acitinib combined with PD-1 mab in the second-line treatment of patients with metastatic renal cancer was significantly higher than that of acitinib (ORR: 33.6% vs. 20.1%, P=0.015) (PFS: 11.7 months vs. 7.5 months, P=0.002).

Piamprilizumab (Anicol) is a new PD-1 monoclonal antibody developed by Zhengda Tianqing Pharmaceutical Group Co., LTD., which has been approved for Hodgkin's lymphoma (R/R cHL) and squamous non-small cell lung cancer (NSCLC) indications in China. Pembrolizumab has achieved significant efficacy in the treatment of classic Hodgkin lymphoma, metastatic nasopharyngeal carcinoma, gastric/esophageal junction adenocarcinoma and other tumor species in clinical studies, with ORR of 89.4%, 29.7% and 26.3%, respectively .

Anicol is a humanized IgG1 subtype of PD-1 monoclonal antibody that eliminates Fc effects. The IgG1 subtype reduces immune escape by eliminating antibody-dependent cell-mediated cytotoxicity (ADCC), antibody-dependent cell-mediated phagocytosis (ADCP), and complement-dependent cytotoxicity (CDC). The combination of anil with FcR can reduce the occurrence of adverse immune reactions , and the incidence of grade 3 and above toxicities such as immune-associated pneumonia, hepatitis, myocardium, and pancreatitis is lower than that of sindillizumab, tirellizumab, and triplizumab. Therefore, this study intends to use anicol combined with anlotinib to explore its efficacy and safety in advanced PPGL.

1.5 Application of antirotinib combined with PD-1 monoclonal antibody in advanced pheochromocytoma/paraganglioma The combination of TKI and PD-1 monoclonal antibody is a research hotspot in the treatment of advanced tumors. Target-free therapy has been widely used in renal, urothelial, lung, liver and other tumors, and has achieved remarkable efficacy [46].

Only a few cases of combined treatment for advanced PPGL have been reported at home and abroad. In Taizhou Hospital of Zhejiang Province in 2022, a patient was treated with palizumab injection 200 mg(once every 3 weeks) for intravenous immunotherapy, combined with anrotinib 10 mg orally (once a day, 14 days and 7 days, every 3 weeks for a course of treatment). The left adrenal mass (9.6cm →8.4cm) and the multiple intrahepatic mass (up to 9.3cm →8.8cm) were both reduced. In the early stage, our team used anrotinib combined with PD-1 monoclonal antibody to treat 3 patients, and the efficacy reached PR 66% (2/3), including 1 case with SHDB mutation. This suggests that targeted immunotherapy for advanced PPGL may have better efficacy.

In an open, multicenter, phase Ib/II clinical study of anlotinib combined with piamprizumab in the treatment of advanced hepatocellular carcinoma, the ORR was 31% and the DCR was 82.8%. The median PFS was 8.8 months (95% CI 4.0-12.3 months). 80% were grade 1/2 toxicity, such as elevated AST, elevated ALT, elevated blood bilirubin, etc. Only 19.4% had grade 3/4 toxicity such as hypertension and rash. This is an improvement in efficacy and a decrease in toxicity compared to the treatment of advanced hepatocellular carcinoma with altilizumab combined with bevacizumab or carrilizumab combined with apatinib.

At present, there have been no studies on the combination of targeted drugs and immunodrugs in the treatment of advanced PPGL at home and abroad. Therefore, this study will for the first time apply the combination of TKI drugs (antirotinib) and PD-1 monoclonal antibody (Pembrolizumab) to metastatic/unresectable pheochromocytoma/paraganglioma, so as to explore the efficacy and safety of combined drugs in the treatment of advanced pheochromocytoma/paraganglioma.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participate in this study and sign informed consent;
* Patients aged ≥18 years and ≤75 years;
* ECOG score ≤2 points; Expected survival ≥6 months;
* Pathological diagnosis of advanced pheochromocytoma/paraganglioma: including clinical stage IV unresectable pheochromocytoma/paraganglioma with postoperative recurrence or metastasis;
* Unwilling or unsuitable for chemotherapy and radionuclide therapy.
* At least one measurable lesion (RECIST 1.1);
* The main organs function well, and the laboratory examination indicators meet:

  1. Blood routine examination:

     Hemoglobin (HB) ≥ 90g/L(5.6 mmol/L); Absolute neutrophil count (ANC) ≥1.5×109/L; Total white blood cells ≥3.5×109/L;

     ③ Platelet (PLT) ≥ 80×109/L;

     Blood biochemical examination:

     ① Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN (liver metastasis/bone metastasis ≤5 × ULN; Bone metastases ≤5 ULN);

     ② Serum total bilirubin (TBIL) ≤1.5 × ULN;

     ③ Serum creatinine Cr≤1.5×ULN or creatinine clearance ≥60 ml/min; Blood urea nitrogen (BUN)≤2.5 × upper limit of normal value (ULN);

     ④ Albumin (ALB)≥30 g/L;
  2. Blood clotting test:

     * Activated partial thromboplastin time (APTT), International standardized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN;
* Women of reproductive age must confirm their non-pregnant status before enrollment, and all enrolled subjects (whether male or female) should take adequate contraceptive measures during the entire treatment period and within 4 weeks after the end of treatment;
* The subjects voluntarily joined the study and were willing to return to the hospital for follow-up, and the compliance was good; Myocardial enzymes and ejection fraction were normal.

Exclusion Criteria:

* known allergic reactions to anrotinib hydrochloride capsules, Benmelstobart active ingredients or any excipients;
* Receiving anti-tumor monoclonal antibodies or other investigational drugs before enrollment; Previous treatment with other anti-PD-1 monoclonal antibodies or other medications targeting PD-1 / PD-L1;
* previous use of anrotinib hydrochloride capsules or other anti-angiogenic drugs, such as Sunitinib, bevacizumab, etc.;
* Patients were taking immunosuppressants or systemic hormone therapy for immunosuppressive purposes (doses greater than 10mg/day prednisone or other equivalent hormones) and were still taking them within 2 weeks prior to enrollment;
* The patient has any active autoimmune disease or a history of autoimmune disease; Have clinical symptoms or diseases of the heart that are not well controlled;
* Congenital or acquired immune deficiency;
* History of gastrointestinal perforation or open biopsy within 4 weeks prior to enrollment; ≥CTCAE grade 3 for any bleeding event, presence of unhealed wounds, ulcers, or fractures;
* Hyperarterial/venous thrombosis events occurred within 6 months before the study period, such as non-cardiovascular and cerebrovascular events (including temporary ischemic attack), deep vein thrombosis (except venous thrombosis caused by intravenous catheterization during previous chemotherapy and cured by investigators), pulmonary embolism, etc.; Cardiac angioplasty or coronary bypass surgery for unstable arrhythmia, unstable angina pectoris or myocardial infarction;
* People with active bleeding or bleeding tendency;
* Correcting QT interval > 480msec; If a patient has QT interval prolongation, but the cause of the prolongation is assessed by the investigator as a pacemaker (and no other cardiac abnormalities), the patient should be considered suitable for inclusion in the study after discussion with the sponsor study physician;
* Patients suspected of having other primary cancers; Patients with other primary malignancies within the 5 years prior to the study (other than adequately treated cervical or skin cancer in situ, such as basal cell carcinoma, squamous cell carcinoma, or non-melanoma skin cancer);
* Combined diseases/medical history:

  1. Clinically significant hemoptysis (> 50ml daily hemoptysis) occurred within 3 months prior to enrollment; Or clinically significant bleeding symptoms or definite bleeding tendencies, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, stool occult blood or above at baseline, or vasculitis;
  2. hypertension, which is not well controlled by antihypertensive drugs (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100mmHg); In the 6 months prior to randomization, the following conditions had occurred: myocardial infarction, severe/unstable angina pectoris, NYHA grade 2 or higher cardiac dysfunction, clinically significant supracentricular or ventricular arrhythmias, and symptomatic congestive heart failure;
  3. interstitial lung disease, non-infectious pneumonia or uncontrollable systemic diseases (such as poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/ L), pulmonary fibrosis and acute pneumonia, etc.); Renal failure requires hemodialysis or peritoneal dialysis; Liver cirrhosis, decompensated liver disease, active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; Hepatitis C, defined as HCV-RNA above the lower detection limit of analytical methods) or chronic hepatitis requiring antiviral therapy;

  (6) Live attenuated vaccine vaccination history within 28 days prior to the first study or live attenuated vaccine vaccination expected during the study period; (7) Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS); Combined with hepatitis B and hepatitis C co-infection; Severe infection, including but not limited to bacteremia requiring hospitalization, severe pneumonia, etc. within 4 weeks before the first dose; Active infection of CTCAE grade ≥2 requiring systemic antibiotic treatment within 2 weeks prior to first administration, or unexplained fever >38.5°C during screening/prior to first administration (fever due to tumor, as determined by the investigator, was eligible for inclusion); Evidence of active tuberculosis infection within 1 year prior to administration; Major surgery within 28 days prior to randomization (tissue biopsy required for diagnosis and insertion of a central venous catheter through peripheral venipentesis [PICC] or infusion PORT is permitted);
* Participants who have previously received or are preparing to receive allogeneic bone marrow transplantation or solid organ transplantation;
* Peripheral neuropathy ≥ grade 2; Patients with active brain metastases, malignant meningitis, spinal cord compression, or imaging CT or MRI findings of brain or pia disease during screening (patients with brain metastases who have completed treatment 14 days before enrollment and whose symptoms are stable can be enrolled, but only after brain MRI, CT or venography evaluation to confirm no symptoms of cerebral hemorrhage);
* significant factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea, and presence of clinically significant intestinal obstruction.
* Women who are pregnant, breastfeeding, planning to become pregnant during the study period, or men or women who are fertile but do not want to use appropriate contraceptive methods.
* The presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participating in the study or interfere with the study results, and patients who are deemed by the investigato
* not suitable for participation in the study;
* Patients with brain metastasis;
* Imaging shows that the tumor has invaded important blood vessels, or follow-up shows that the tumor is highly likely to invade important blood vessels and cause fatal bleeding;
* Drugs that interact with anlotinib hydrochloride capsules/piamplizumab are being used;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2years
  The sum of the maximum tumor diameter decreased by ≥30%

SECONDARY OUTCOMES:
progression-free survival | 2years
  The time before tumor diameters increased by less than 20%
Overall survival | 2years
  The time before the patient died
Duration of remission | 2years
  The duration of tumor remission
Clinical response rate | 2years
  the number of patient with PR SD and CR

CONTACTS AND LOCATIONS:
Overall Officials: Shengjie Guo, Doctor, Study Chair — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China